CLINICAL TRIAL: NCT02575261
Title: Chimeric Antigen Receptor-Modified T Cells for EphA2 Positive Recurrent and Metastatic Malignant Glioma
Brief Title: CAR-T Cell Immunotherapy for EphA2 Positive Malignant Glioma Patients
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fuda Cancer Hospital, Guangzhou (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAR-T for malignant glioma
Record Dates: First submitted 2015-09-29; First posted 2015-10-14 (Estimated); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: EphA2 Positive Malignant Glioma; CAR-T Cell Immunotherapy
Keywords: CAR-T cell immunotherapy; EphA2; malignant glioma
MeSH Terms: conditions — Glioma | interventions — Immunotherapy, Adoptive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental:CAR-T cell immunotherapy (Experimental): Enrolled patients will receive CAR-T cell immunotherapy with a novel specific Chimeric antigen receptor aiming at EphA2 antigen by infusion.
  Interventions: Biological: CAR-T cell immunotherapy
- No Intervention (No Intervention)

INTERVENTIONS:
Biological: CAR-T cell immunotherapy — This CAR-T cell immunotherapy with a novel specific Chimeric antigen receptor aiming at EphA2 antigen.
  Arms: Experimental:CAR-T cell immunotherapy

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of CAR-T cell immunotherapy in treating with EphA2 positive malignant glioma patients.

DETAILED DESCRIPTION:
Chimeric antigen receptor (CAR) is a recombinant receptor with both antigen-binding and T cell activating functions. Chimeric antigen receptor T cell Immunotherapy has more advantages compared with conventional immunotherapy, especially in dealing with patients of hematologic malignancies and solid malignant tumors.This study design a novel specific Chimeric antigen receptor aiming at EphA2 antigen.After CAR-T cell infusion,At periodic intervals, the investigators will evaluate clinical symptoms Improved conditions of this disease.Through this study,the investigators will evaluate the safty and effectiveness of CAR-T cell immunotherapy in treating with EphA2 positive malignant glioma patients.

ELIGIBILITY:
Inclusion Criteria:

1. the primary EphA2 positive patients, the best are malignant glioma patients.
2. the recurrent EphA2 positive patients, the best are malignant glioma patients.
3. Patients must have evidence of adequate bone marrow reserve, hepatic and renal function as evidenced by the following laboratory parameters:

Absolute neutrophil count greater than 1500/mm3. Platelet count greater than 100,000/mm3. Hemoglobin greater than 10g/dl (patients may receive transfusions to meet this parameter).

Total bilirubin < 1.5 times upper limits of normal. Serum creatinine less than or equal to 1.6 mg/ml or the creatinine clearance must be greater than 70 ml/min/1.73m(2).

* Seronegative for HIV antibody.
* Seronegative for active hepatitis B, and seronegative for hepatitis C antibody.
* Patients must be willing to practice birth control during and for four months following treatment.NOTE:women of child-bearing age must have evidence of negative pregnancy test.
* Patients must be willing to sign an informed consent.

Exclusion Criteria:

1. the patients with multiple kinds of cancars are excluded.
2. Patients with uncontrolled hypertension (> 160/95), unstable coronary disease evidenced by uncontrolled arrhythmias, unstable angina, decompensated congestive heart failure (> New York Heart Association Class II), or myocardial infarction within 6 months of study will be excluded.
3. Patients with any of the follo wing pulmonary function abnormalities will be excluded: FEV(forced expiratory volume), < 30% predicted; DLCO (diffusing capacity of lung for carbon monoxide) < 30% predicted (post-bronchodilator); Oxygen Saturation less than 90% on room air.
4. Patients with severe liver and kidney dysfunction or consciousness disorders will be excluded.
5. Pregnant and/or lactating women will be excluded.
6. Patients with active infections, including HIV, will be excluded, due to unknown effects of the vaccine on lymphoid precursors.
7. Patients with any type of primary immunodeficiencies will be excluded from the study.
8. Patients requiring corticosteroids (other than inhaled) will be excluded.
9. Patients with history of T cell tumors will be excluded.
10. Patients who are participating or participated any other clinical trials in latest 30 days will be excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2016-08-15 (Actual); Study Completion 2016-08-15 (Actual)

PRIMARY OUTCOMES:
The effectiveness of CAR-T cell immunotherapy | 24 weeks
  After CAR-T cell infusion,we will detect the persistence of CAR-T cells by flow-cytometric analysis.And we will observe if this CAR T cells can significantly inhibite the tumor growth by discovering the change of tumor volume.

SECONDARY OUTCOMES:
The safety of CAR-T cell immunotherapy (adverse events) | 6 weeks
  After CAR-T cell infusion,we will observe the potential adverse events related to the T-cell infusion such as high fever,jaundice, kidney failure and so on.

OTHER OUTCOMES:
Clinical response | 24 weeks
  Clinical response to T-cell infusion, especially change of tumor volume will be evaluated by comparing disease identified by computed tomography, magnetic resonance imaging, and/or positron emission tomography images.
Progress free disease (PFS) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Lizhi Niu, PhD, Study Chair — Fuda Cancer Hospital
Locations (1):
- Central laboratory in Fuda cancer hospital, Guangzhou, Guangdong, China